CLINICAL TRIAL: NCT02907866
Title: Use of Endobronchial Ultrasound Scope (EBUS) Transducer to Identify Pneumothorax-A Feasibility Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: 6622
Record Dates: First submitted 2016-09-14; First posted 2016-09-20 (Estimated); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Pneumothorax
MeSH Terms: conditions — Pneumothorax | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Patients undergoing bronchoscopy: All patients presenting for bronchoscopy (These patient are expected to have normal pleural sliding sign identified by ultrasound)
  Interventions: Device: Ultrasound with EBUS scope and with linear ultrasound probe
- Patients with pneumothorax: Patients with pneumothorax requiring chest tube(This group of patient is expected to have residual pneumothorax for identification of absence of lung sliding, B lines and lung point)
  Interventions: Device: Ultrasound with EBUS scope and with linear ultrasound probe
- Patients on mechanical ventilation: Patients with respiratory failure on mechanical ventilation(This group of patient is expected to have alveolo-interstitial findings such as B lines)
  Interventions: Device: Ultrasound with EBUS scope and with linear ultrasound probe

INTERVENTIONS:
Device: Ultrasound with EBUS scope and with linear ultrasound probe — All subjects will have an ultrasound of the chest performed with the tip of the EBUS scope as well as the linear ultrasound probe, which will be used as a reference for comparison. At the end of the procedure, while the patient in the supine position, the transducer of the EBUS bronchoscope will be placed on the anterior thorax, superficial to the skin and in a sagittal direction that is perpendicular to 2 ribs. The depth of the ultrasound beam will be increased to identify the pleural sliding sign and B lines (vertical lines) when present.This will be followed by use of linear ultrasound probe to scan the chest wall for normal lung sliding, B-lines and potential pneumothorax. The patient will remain in supine position. The linear probe will be placed on anterior thorax at the level of second intercostal space. The depth of the ultrasound beam will be adjusted to identify lung sliding and B-lines.

SUMMARY:
Endobronchial ultrasound (EBUS) is a technique that uses ultrasound along with bronchoscope to visualize airway wall and structures adjacent to it. Pneumothorax is a known complication from EBUS procedure. To rule out a Pneumothorax after the procedure, a Chest -X-ray is usually done. Point-of-care sonography has emerged as an invaluable tool in the assessment of patients with both traumatic and non-traumatic dyspnea. Multiple studies involving bedside ultrasound has shown that a pneumothorax can easily be ruled out if pleural sliding sign or B lines are visualized on lung ultrasonography; the accuracy of lung ultrasound in ruling out pneumothorax approach computed tomography and exceed plain radiography. Preforming a lung ultrasound using the EBUS bronchoscope tip as a way to rule out pneumothorax has never been described previously. If this is possible it will obviate the need of getting a Chest -X-ray and decrease the dose of radiation that the patient is exposed to. In this study we will demonstrate that the feasibility of using the transducer of the EBUS Bronchoscope to perform bedside lung ultrasound to rule out pneumothorax.

DETAILED DESCRIPTION:
The use of ultrasound in diagnosis and treatment of patients has been well-established for many decades. The use of thoracic ultrasonography is a fairly new and rapidly evolving field. The interface between the ultrasound probe and chest wall can produce artifacts that can be useful in diagnosing a pneumothorax. In one prospective study the utility of ultrasound was compared to chest X-ray and CT-scan by trauma surgeon (1). Their results demonstrate that ultrasound was more sensitive than chest X-ray to identify early pneumothorax. The study also demonstrated that 63% of pneumothoraxes diagnosed were occult and would have been later diagnosed on CT chest. In these critical situations where is subtle pneumothorax can be missed, a bedside ultrasound has been proven to accelerate the diagnosis and thus treatment. Similarly another prospective study noted that up to 76% of all traumatic pneumothoraxes were missed by standard AP chest X-ray, when interpreted by trauma team (2). This number was significantly higher than a retrospective study in which 55% of pneumothoraxes were missed on AP chest films reviewed by radiologist (3). The sensitivity of ultrasound in detecting pneumothorax has been demonstrated in multiple studies to be similar to CT-scan, which is considered to be gold standard for the detection of pneumothorax (4, 5).

Visualization of normal pleural lung sliding is itself sufficient to exclude pneumothorax , if lung sliding is not present the finding of B lines( vertical lines), which usually originate from the lung parenchyma will also exclude the possibility of pneumothorax at the interspace in question, since the lung parenchyma cannot be visualized if there is air interposed between the pleura and the lung.

Endobronchial ultrasound (EBUS) is considered an integral component of diagnosis of indeterminate mediastinal lymph nodes, masses and peripheral pulmonary nodules. EBUS is minimally invasive, safe and highly accurate (6). According to current estimates that incidence if complications associated with EBUS is between 1-1.5% (6, 7). Major complications are associated with needle aspirations. The incidence of pneumothorax was found to be 3.3% in one retrospective analysis (8), with 31% of patients requiring chest tube eventually for treatment of pneumothorax. Post-procedure chest-X-rays are commonly performed to rule out pneumothorax. Based on current data chest-X-rays are considered suboptimal for diagnosis of pneumothorax and can also expose patients to undue radiation.

The EBUS probe contains a small ultrasound through which ultrasound images of various structure i.e. lymph nodes, ventricles, pulmonary vasculature can be visualized. Ruling out pneumothorax via lung ultrasound using EBUS probe has never been described. If this is possible, it avoids the need of obtaining post-procedure Chest-X-rays thus decreasing the dose of radiation exposure and prevent time delays for the arrival of chest-x-rays.

In this study we will demonstrate the feasibility of using the transducer of the EBUS Bronchoscope to perform bedside lung ultrasound to rule out pneumothorax.

ELIGIBILITY:
Inclusion Criteria:

1. All patients presenting for bronchoscopy (These patient are expected to have normal pleural sliding sign identified by ultrasound)
2. Patients with pneumothorax requiring chest tube(This group of patient is expected to have residual pneumothorax for identification of absence of lung sliding, B lines and lung point)
3. Patients with respiratory failure on mechanical ventilation(This group of patient is expected to have alveolo-interstitial findings such as B lines)

Exclusion Criteria:

-Absence of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. All patients presenting for bronchoscopy (These patient are expected to have normal pleural sliding sign identified by ultrasound)
  2. Patients with pneumothorax requiring chest tube(This group of patient is expected to have residual pneumothorax for identification of absence of lung sliding, B lines and lung point)
  3. Patients with respiratory failure on mechanical ventilation(This group of patient is expected to have alveolo-interstitial findings such as B lines)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients on whom a sliding sign and/or B lines are identified successfully with EBUS versus linear US | 1 Hour

SECONDARY OUTCOMES:
Sensitivity, specificity, negative and positive predictive value of the bedside lung ultrasound using the EBUS transducer to detect pneumothorax as compared to the linear US, the bedside Chest X-ray and the final clinical diagnosis of pneumothorax. | 1 Hour
The Time elapsed between the end of the bronchoscopy and the completion of lung ultrasound will be compared to the time between the end of the bronchoscopy and the availability of CXR imaging. | 1 Hour

CONTACTS AND LOCATIONS:
Locations (1):
- Oklahoma University Medical center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kirkpatrick AW, Sirois M, Laupland KB, Liu D, Rowan K, Ball CG, Hameed SM, Brown R, Simons R, Dulchavsky SA, Hamiilton DR, Nicolaou S. Hand-held thoracic sonography for detecting post-traumatic pneumothoraces: the Extended Focused Assessment with Sonography for Trauma (EFAST). J Trauma. 2004 Aug;57(2):288-95. doi: 10.1097/01.ta.0000133565.88871.e4. PMID 15345974
- [Background] Ball CG, Ranson K, Dente CJ, Feliciano DV, Laupland KB, Dyer D, Inaba K, Trottier V, Datta I, Kirkpatrick AW. Clinical predictors of occult pneumothoraces in severely injured blunt polytrauma patients: A prospective observational study. Injury. 2009 Jan;40(1):44-7. doi: 10.1016/j.injury.2008.07.015. Epub 2009 Jan 8. PMID 19131061
- [Background] Ball CG, Kirkpatrick AW, Laupland KB, Fox DI, Nicolaou S, Anderson IB, Hameed SM, Kortbeek JB, Mulloy RR, Litvinchuk S, Boulanger BR. Incidence, risk factors, and outcomes for occult pneumothoraces in victims of major trauma. J Trauma. 2005 Oct;59(4):917-24; discussion 924-5. doi: 10.1097/01.ta.0000174663.46453.86. PMID 16374282
- [Background] Blaivas M, Lyon M, Duggal S. A prospective comparison of supine chest radiography and bedside ultrasound for the diagnosis of traumatic pneumothorax. Acad Emerg Med. 2005 Sep;12(9):844-9. doi: 10.1197/j.aem.2005.05.005. PMID 16141018
- [Background] Soldati G, Testa A, Sher S, Pignataro G, La Sala M, Silveri NG. Occult traumatic pneumothorax: diagnostic accuracy of lung ultrasonography in the emergency department. Chest. 2008 Jan;133(1):204-11. doi: 10.1378/chest.07-1595. Epub 2007 Oct 9. PMID 17925411
- [Background] Asano F, Aoe M, Ohsaki Y, Okada Y, Sasada S, Sato S, Suzuki E, Semba H, Fukuoka K, Fujino S, Ohmori K. Complications associated with endobronchial ultrasound-guided transbronchial needle aspiration: a nationwide survey by the Japan Society for Respiratory Endoscopy. Respir Res. 2013 May 10;14(1):50. doi: 10.1186/1465-9921-14-50. PMID 23663438
- [Background] Eapen GA, Shah AM, Lei X, Jimenez CA, Morice RC, Yarmus L, Filner J, Ray C, Michaud G, Greenhill SR, Sarkiss M, Casal R, Rice D, Ost DE; American College of Chest Physicians Quality Improvement Registry, Education, and Evaluation (AQuIRE) Participants. Complications, consequences, and practice patterns of endobronchial ultrasound-guided transbronchial needle aspiration: Results of the AQuIRE registry. Chest. 2013 Apr;143(4):1044-1053. doi: 10.1378/chest.12-0350. PMID 23117878
- [Background] Huang CT, Ruan SY, Liao WY, Kuo YW, Lin CY, Tsai YJ, Ho CC, Yu CJ. Risk factors of pneumothorax after endobronchial ultrasound-guided transbronchial biopsy for peripheral lung lesions. PLoS One. 2012;7(11):e49125. doi: 10.1371/journal.pone.0049125. Epub 2012 Nov 7. PMID 23145094